CLINICAL TRIAL: NCT03816085
Title: The Effects of Shoes With Different Heel Heights on Balance, Muscular Endurance and Functional Skills
Brief Title: Shoes on Balance, Muscular Endurance and Functional Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ETK00-2018-0239
Record Dates: First submitted 2019-01-02; First posted 2019-01-25 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: women; shoes; balance; muscles
MeSH Terms: interventions — Shoes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Shoe with 4 cm heel (Experimental): Shoes with 4 cm heel will be applied to women. Tests to measure balance, muscular endurance and function will be done while they wear this shoe.
  Interventions: Other: Shoes
- Shoe with 10 cm heel (Experimental): Shoes with 10 cm heel will be applied to women. Tests to measure balance, muscular endurance and function will be done while they wear this shoe.
  Interventions: Other: Shoes
- Without shoes (No Intervention): Women will be included in the tests to measure balance, muscular endurance and function without shoes.

INTERVENTIONS:
Other: Shoes — Shoes with different heel heights
  Other Names: Women wearing shoes
  Arms: Shoe with 10 cm heel; Shoe with 4 cm heel

SUMMARY:
In daily life, stiletto heeled shoes which are popularly preferred by women have different heel heights. This study aims to investigate the effects of these differences on balance, muscular endurance and functional skills. Heel heights were chosen as 4 and 10 cm. Other features of shoes (stiletto type/colour etc.) will be same. The tests will be randomly done barefoot, 10 cm, and 4cm shoes.

DETAILED DESCRIPTION:
The evaluations will include Functional Forward Reach Test for dynamic balance and Single Leg Standing for static balance, heel raising and squat-up test for muscular endurance of plantar flexor and quadriceps muscles, ascending stairs for functional skills.

Measuring distance will be used for Functional reach test and timing will be used for single leg standing test. Timing and repetition number will be used for muscular endurance tests. Timing will be used to climb up 10 stairs with and without heel contact.

ELIGIBILITY:
Inclusion Criteria:

* the shoe number will be 37
* women who do not regularly wear high heeled shoes
* women who are familiar with stiletto heeled shoes

Exclusion Criteria:

* any pain which prevents to participate in tests
* women with cardiovascular disease, metabolic disease, blood pressure disorders, diabetes diseases, neuromuscular diseases.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Heeled shoes are used among women.
Enrollment: 40 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Functional Skill | at baseline
  The case will be asked to climb up 10 stairs as fast as possible. Time (in seconds) will be recorded for climbing up with and without heel contact.

SECONDARY OUTCOMES:
Single Leg Standing | at baseline
  The case will be asked to stand on dominant leg. If the raised leg touches anything around (other limb, floor) or in condition of hopping/splashing, time will be stopped. Time (seconds) will be recorded.

OTHER OUTCOMES:
Repetition number of heel raising | at baseline
  Before the test, the case will be asked to stretch plantar flexor muscles. Then the case will be asked to raise the heels unilaterally. The repetition number will be written until the case cannot do the full movement.
Repetition number of squating | at baseline
  Before the test, the case will be asked to stretch quadriceps muscle with flexing the knee. Then the case will be asked to squat continuously. The repetition number will be written until the case cannot do the full movement.
Duration of heel raising | at baseline
  Before the test, the case will be asked to stretch plantar flexor muscles. Then the case will be asked to raise the heels unilaterally. The time (in seconds) will be written until the case cannot do the full movement.
Duration of squating | Before the test, the case will be asked to stretch quadriceps muscle with flexing the knee. Then the case will be asked to squat continuously. The repetition number will be written until the case cannot do the full movement.
  Before the test, the case will be asked to stretch quadriceps muscle with flexing the knee. Then the case will be asked to squat continuously. The time (in seconds) will be written until the case cannot do the full movement.
Functional Forward Reach Test | Before the test, the case will be asked to stretch quadriceps muscle with flexing the knee. Then the case will be asked to squat continuously. The repetition number will be written until the case cannot do the full movement.
  Before the test, the case will be asked to stretch quadriceps muscle with flexing the knee. Then the case will be asked to squat continuously. The repetition number will be written until the case cannot do the full movement.

CONTACTS AND LOCATIONS:
Overall Officials: ZEHRA GÜÇHAN TOPCU, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Zehra Güçhan Topcu, Famagusta, Cyprus